CLINICAL TRIAL: NCT02482519
Title: The Effects of Acute Weight Gain and Acute Calorie Deprivation on Marrow Adipose Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Chief, Neuroendocrine Unit, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015P000624
Record Dates: First submitted 2015-06-16; First posted 2015-06-26 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Healthy
MeSH Terms: interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 10 day overfeeding/fasting (Other): 10 day high calorie diet followed by a 10 day fast
  Interventions: Other: High calorie diet; Other: Fasting

INTERVENTIONS:
Other: High calorie diet — High calorie diet for 10 days
Other: Fasting — 10 day fast

SUMMARY:
Marrow adipocytes have been identified as a component of the bone marrow micro-environment. Evidence exists suggesting that marrow fat plays an important physiologic role in both bone mineral and energy metabolism in humans. The investigators will study the effects of acute weight gain and acute nutritional deprivation on energy homeostasis and bone mineral metabolism by examining marrow adiposity, peripheral fat depots and bone microarchitecture.

The study will include two ten day inpatient study visits. Participants will eat a high calorie diet for 10 days, followed by a 13-18 day stabilization period at home, and then return for a ten day fast.

DETAILED DESCRIPTION:
Marrow adipocytes have been identified as a component of the bone marrow micro-environment. Evidence exists suggesting that marrow fat plays an important physiologic role in both bone mineral and energy metabolism in humans. Studies have shown that nutritional status, particularly body fat distribution, may be important in marrow fat. For example, anorexia nervosa, a state of low body fat, is associated with elevated marrow adiposity and low bone mineral density. However, it is not known whether this is in direct response to nutritional deprivation or other hormonal changes that occur in anorexia nervosa. Drugs known to cause adipose redistribution and associated with low bone mass, such as the thiazolidinediones and glucocorticoids, have also been shown to stimulate the accumulation of marrow adipocytes. Therefore, the relationship between bone marrow fat, bone mass, body fat depots and their hormone regulators is a dynamic one and not yet well understood. Although studies have shown an inverse relationship between high marrow adiposity and low bone mineral density (BMD), the physiologic role of marrow adipose tissue has not been defined nor its relationship to hormonal factors in humans. A role for marrow adipose tissue (MAT) in mineral and energy metabolism is further supported by the fact that a number of pathologic states are associated with increased marrow adiposity. Visceral adipose tissue, intramyocellular lipids (IMCL), intrahepatic lipids (IHL) and serum triglycerides, all of which are elevated in obesity, are also positive predictors of MAT, but whether acute weight gain in humans results in elevated marrow adiposity is unknown. Therefore observing changes in marrow fat during acute weight gain and acute nutritional deprivation will further the understanding of the role of marrow adiposity in energy homeostasis. While it is known that markers of bone formation dramatically decrease after only 4 days of fasting, it is not known how quickly marrow fat can change in response to physiologic cues. In a rat model, increases in marrow fat were observed after 14 days in space suggesting that changes in marrow adiposity may occur acutely in the human model as well.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, ages 21-45 years
2. 101-120% of ideal body weight as defined by the 1983 Metropolitan Life Insurance Height and Weight Tables
3. Normal thyroid function
4. Regular menses (women) - Female subjects will start the study within 1 week of Day 1 of their menstrual period
5. Normal transaminase levels (AST/ALT)

Exclusion Criteria:

1. Any disease known to affect bone metabolism, including untreated thyroid dysfunction, Cushing's syndrome, or renal failure
2. Any medication known to affect bone metabolism -- including systemic steroids or immunosuppressants -- within three months of the study, excluding estrogen and progestins. Patients receiving depot medroxyprogesterone (Depo-Provera) will be excluded from participating for six months after their last injections. Bisphosphonates must have been discontinued for at least one year before participation
3. Serum potassium <3.0 meq/L
4. History of eating disorder
5. Pregnant and/or breastfeeding (women)
6. Diabetes mellitus
7. Active substance abuse, including alcohol
8. Contraindications to MRI: cardiac pacemaker, metal implants, claustrophobia
9. History of chemotherapy or radiation therapy
10. History of a bleeding disorder or use of anti-platelet medications
11. Allergy to allopurinol
12. The study physician feels that the subject may not be able to safely complete the study or may place themselves at risk by undergoing the study

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-11; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Marrow adiposity will be measured using magnetic resonance spectroscopy | Change from baseline marrow adipose tissue after high-calorie diet and after fast (35 days)
  Marrow adipose tissue measurement of the spine and hip

CONTACTS AND LOCATIONS:
Overall Officials: Anne Klibanski, MD, Principal Investigator — MGH/Harvard Medical School
Locations (1):
- Massachusettes General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Colling C, Bredella MA, Fazeli PK, Pachon-Pena G, Singh RJ, Rosen CJ, Miller KK. Changes in serum cortisol levels after 10 days of overfeeding and fasting. Am J Physiol Endocrinol Metab. 2023 Jun 1;324(6):E506-E513. doi: 10.1152/ajpendo.00181.2022. Epub 2023 Apr 13. PMID 37053050